CLINICAL TRIAL: NCT03323749
Title: A Phase 3 Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Daily Subcutaneous Injections of Elamipretide in Subjects With Primary Mitochondrial Myopathy Followed by an Open-Label Treatment Extension
Brief Title: A Trial to Evaluate Safety and Efficacy of Elamipretide Primary Mitochondrial Myopathy Followed by Open-Label Extension
Acronym: MMPOWER-3
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Part1,double blind portion of the trial did not meet the primary end points
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIMM-301
Record Dates: First submitted 2017-10-12; First posted 2017-10-27 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Primary Mitochondrial Myopathy
Keywords: Myopathy; PMD; Primary Mitochondrial Disease; MTP-131; elamipretide
MeSH Terms: conditions — Muscular Diseases | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Elamipretide (Experimental): 40 mg (0.5mL) elamipretide subcutaneous (SC) daily
  Interventions: Combination Product: elamipretide
- Part 1: Placebo (Placebo Comparator): Placebo SC daily
  Interventions: Combination Product: placebo comparator
- Part 2: Elamipretide open label (Experimental): Elamepretide 40 mg (0.5 mL) SC daily
  Interventions: Combination Product: elamipretide open label treatment

INTERVENTIONS:
Combination Product: elamipretide — 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system
  Other Names: MTP-131
  Arms: Part 1: Elamipretide
Combination Product: placebo comparator — 40 mg of placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system
  Other Names: Placebo
  Arms: Part 1: Placebo
Combination Product: elamipretide open label treatment — 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
  Arms: Part 2: Elamipretide open label

SUMMARY:
This is a multicenter phase 3 randomized, double-blind, parallel-group, placebo-controlled trial to evaluate the safety and efficacy of daily subcutaneous injections of elamipretide in subjects with primary mitochondrial myopathy. This will be followed by an open-label treatment extension.

DETAILED DESCRIPTION:
Part 11 is a 24-week, randomized, double-blind, parallel-group, placebo-controlled assessment of the efficacy and safety of single daily subcutaneous (SC) doses of 40 mg elamipretide (vs placebo) administered with the elamipretide delivery system as a treatment for subjects with primary mitochondrial myopathy (PMM). Part 2 was to assess the long-term safety and tolerability of single daily SC doses of 40 mg elamipretide administered with the elamipretide delivery system for up to 144 weeks.

ELIGIBILITY:
PART 1:

Inclusion Criteria:

* Willing and able to provide a signed informed consent form prior to participation in any trial-related procedures
* Agrees to adhere to the trial requirements for the length of the trial, including the use of the elamipretide delivery system
* Subject is ≥ 16 and ≤ 80 years of age
* Diagnosed with PMM in the opinion of the investigator and confirmed by an Adjudication Committee
* Woman of childbearing potential must agree to use a highly effective method of birth control

Exclusion Criteria:

* Subject has myopathic signs and or/symptoms due to a neuropathic process or gait problem that would interfere with the 6 minute walk test (6MWT), in the opinion of the Investigator
* Female who are pregnant, planning to become pregnant, or breastfeeding/lactating
* At Screening, the estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m^2
* Subject has undergone an in-patient hospitalization within the 30 days prior to the Baseline Visit or has a planned hospitalization or a surgical procedure during the trial.
* Subject has clinically significant cardiac disease or prior interventional procedure and/or respiratory disease (medical history or current clinical findings) within 3 months of the Baseline Visit, in the opinion of the Investigator.
* Subject has QTc elongation (using the correction factor utilized at the clinical site) defined as a QTc >450 msec in male subjects and >480 msec in female subjects.
* ECG evidence of acute ischemia, atrial fibrillation, or active conduction system abnormalities with the exception of any of the following:

  1. First degree Atrioventricular bock (AV-block)
  2. Second degree AV-block Type 1 (Mobitz Type 1 / Wenckebach type)
  3. Right bundle branch block
* Subject has severe vision impairment that, in the opinion of the Investigator, may interfere with their ability to complete all trial requirements
* Subject has a seizure disorder that, in the opinion of the Investigator, may interfere with their ability to complete all trial requirements.
* Active malignancy or any other cancer from which the subject has been disease-free for < 2 years.
* Subject has a solid organ transplant and/or is currently receiving treatment with therapy for immunosuppression, in the opinion of the Investigator.
* Subject has been previously diagnosed with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
* Subject has a history of a systemic eosinophilic illness and/or an eosinophil count >1,000 cells x10^6/L at the Screening Visit.
* Subject is currently participating or has participated in an interventional clinical trial (i.e.,investigational product or device, stem cell therapy, gene therapy) within 30 days of the Baseline Visit; or is currently enrolled in a non-interventional clinical trial (except for SPIMM-300) at the Baseline Visit which, in the opinion of the Investigator, may be potentially confounding with results of the current trial (e.g., exercise therapy trial).
* Subject has previously received elamipretide (MTP-131), for any reason.
* Subject has a history of active substance abuse during the year before the Baseline Visit, in the opinion of the Investigator.
* Subject has any prior or current medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all trial requirements.

PART 2:

Continuation Criteria:

* Subjects must continue to be able and willing to adhere to the trial requirements.
* Subject is appropriate to continue in Part 2 (i.e. subject was compliant in Part 1), in the opinion of the Investigator.
* Subject has not had a serious adverse event (SAE)/serious adverse device effect (SADE) attributed to the elamipretide delivery system.
* Subject has not permanently discontinued the elamipretide delivery system.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (13):
  - University of California San Diego, La Jolla, California
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rare Disease Research, LLC, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinical Neurological Institute, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine/Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - Adult Metabolic Diseases Clinic, Vancouver, British Colombia
  - McMaster University Medical Center, Hamilton, Ontario
- Copenhagen Neuromuscular Center, Copenhagen, Denmark
- Germany (2):
  - University Hospital of Bonn, Bonn
  - Klinikum der Universität München, Friedrich-Baur Institute, Munich
- Institute of Genomic Medicine and Rare Disorders, Budapest, Hungary
- Italy (6):
  - IRCCS Institute of Neorological Sciences of Bologna, Bellaria Hospital, Bologna
  - Azienda Ospedaliero Universitaria Policlinico G. Martino, Messina
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Dipartimento Ambientale di Neuroscienze, Pisa
  - Ospedale Pediatrico Bambin Gesù, Rome
  - Istituto di Neurologia, Fondazione Policlinico Universitario A. Gemelli, Rome
- United Kingdom (2):
  - MRC Centre for Neuromuscular Diseases, London
  - Royal Victoria Infirmary, Newcastle upon Tyne

REFERENCES:
- [Derived] Karaa A, Bertini E, Carelli V, Cohen B, Ennes GM, Falk MJ, Goldstein A, Gorman G, Haas R, Hirano M, Klopstock T, Koenig MK, Kornblum C, Lamperti C, Lehman A, Longo N, Molnar MJ, Parikh S, Phan H, Pitceathly RDS, Saneto R, Scaglia F, Servidei S, Tarnopolsky M, Toscano A, Van Hove JLK, Vissing J, Vockley J, Finman JS, Abbruscato A, Brown DA, Sullivan A, Shiffer JA, Mancuso M; MMPOWER-3 Trial Investigators. Genotype-specific effects of elamipretide in patients with primary mitochondrial myopathy: a post hoc analysis of the MMPOWER-3 trial. Orphanet J Rare Dis. 2024 Nov 21;19(1):431. doi: 10.1186/s13023-024-03421-5. PMID 39574155
- [Derived] Karaa A, Bertini E, Carelli V, Cohen BH, Enns GM, Falk MJ, Goldstein A, Gorman GS, Haas R, Hirano M, Klopstock T, Koenig MK, Kornblum C, Lamperti C, Lehman A, Longo N, Molnar MJ, Parikh S, Phan H, Pitceathly RDS, Saneto R, Scaglia F, Servidei S, Tarnopolsky M, Toscano A, Van Hove JLK, Vissing J, Vockley J, Finman JS, Brown DA, Shiffer JA, Mancuso M; MMPOWER-3 Trial Investigators. Efficacy and Safety of Elamipretide in Individuals With Primary Mitochondrial Myopathy: The MMPOWER-3 Randomized Clinical Trial. Neurology. 2023 Jul 18;101(3):e238-e252. doi: 10.1212/WNL.0000000000207402. Epub 2023 Jun 2. PMID 37268435

RESULTS

PARTICIPANT FLOW:
Groups:
- Double-Blind Elamipretide, Then Open Label Elamepretide: 40 mg (0.5mL) elamipretide subcutaneous (SC) daily
  elamipretide: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system, then elamipretide open-label treatment: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
- Double-Blind Placebo Then Open-Label Elamepretide: Placebo SC daily
  Double-blind period: placebo comparator: Placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system. Open-label period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system.
Period: Double-blind Period
Arm/Group | Double-Blind Elamipretide, Then Open Label Elamepretide | Double-Blind Placebo Then Open-Label Elamepretide
Started | 109 | 109
Completed | 102 | 103
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 4 | 5
Not completed — Adverse Event | 3 | 1
Period: Open-Label Period
Arm/Group | Double-Blind Elamipretide, Then Open Label Elamepretide | Double-Blind Placebo Then Open-Label Elamepretide
Started (A total of 196 subjects enrolled in Part 2 of the trial: 93 from the elamipretide group in Part 1, and 103 from the placebo group in Part 1. No subjects completed the trial: it was terminated early due to the Sponsor's decision.) | 93 | 103
Completed | 0 | 0
Not Completed | 93 | 103
Not completed — Termination of the Clinical Development of Elamipretide in Subjects with PMM | 83 | 88
Not completed — Adverse Event | 3 | 10
Not completed — Withdrawal by Subject | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Elamipretide: Double-blind Period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system, then Open-label Period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
- Placebo: Double-Blind Period: Placebo comparator: 40 mg of placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks, then Open-label Period: Elamipretide: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
- Total: Total of all reporting groups
Arm/Group | Elamipretide | Placebo | Total
Number analyzed (Participants) | 109 | 109 | 218
Age, Customized [Mean (Standard Deviation); unit: years] — Population: Open-label Period: A total of 196 Subjects enrolled in the Open-Label Extension: 93 from the original Double-Blind Period Elamipretide group and 103 from the original Double-Blind Placebo group.
  years
    Years, Double-blind | 45.5 (15.72) | 44.3 (14.34) | 44.9 (15.02)
    Years, Open-label: number analyzed (Participants) | 93 | 103 | 196
    Years, Open-label | 45.7 (15.97) | 45.0 (14.25) | 45.3 (15.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Open-label Period: A total of 196 Subjects enrolled in the Open-Label Extension: 93 from the original Double-Blind Period Elamipretide group and 103 from the original Double-Blind Placebo group.
  Participants
    Double-Blind Sex: Female | 67 | 73 | 140
    Double-Blind Sex: Male | 42 | 36 | 78
    Open-Enrollment Sex: number analyzed (Participants) | 93 | 103 | 196
    Open-Enrollment Sex: Female | 56 | 67 | 123
    Open-Enrollment Sex: Male | 37 | 36 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Open-label Period: A total of 196 Subjects enrolled in the Open-Label Extension: 93 from the original Double-Blind Period Elamipretide group and 103 from the original Double-Blind Placebo group.
  Participants
    Ethnicity Double-Blind: Hispanic or Latino | 11 | 10 | 21
    Ethnicity Double-Blind: Not Hispanic or Latino | 95 | 96 | 191
    Ethnicity Double-Blind: Unknown or Not Reported | 3 | 3 | 6
    Ethnicity Open-Label: number analyzed (Participants) | 93 | 103 | 196
    Ethnicity Open-Label: Hispanic or Latino | 8 | 10 | 18
    Ethnicity Open-Label: Not Hispanic or Latino | 82 | 91 | 173
    Ethnicity Open-Label: Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Open-label Period: A total of 196 Subjects enrolled in the Open-Label Extension: 93 from the original Double-Blind Period Elamipretide group and 103 from the original Double-Blind Placebo group.
  Participants
    Double-blind Period: American Indian or Alaska Native | 1 | 0 | 1
    Double-blind Period: Asian | 2 | 5 | 7
    Double-blind Period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Double-blind Period: Black or African American | 1 | 0 | 1
    Double-blind Period: White | 103 | 100 | 203
    Double-blind Period: More than one race | 2 | 1 | 3
    Double-blind Period: Unknown or Not Reported | 0 | 3 | 3
    Open-label period: number analyzed (Participants) | 93 | 103 | 196
    Open-label period: American Indian or Alaska Native | 1 | 0 | 1
    Open-label period: Asian | 0 | 4 | 4
    Open-label period: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Open-label period: Black or African American | 1 | 0 | 1
    Open-label period: White | 89 | 95 | 184
    Open-label period: More than one race | 2 | 1 | 3
    Open-label period: Unknown or Not Reported | 0 | 3 | 3
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: Open-label Period: A total of 196 Subjects enrolled in the Open-Label Extension: 93 from the original Double-Blind Period Elamipretide group and 103 from the original Double-Blind Placebo group.
  kg
    Double-blind | 64.81 (20.287) | 67.24 (17.336) | 66.02 (18.865)
    Open-label: number analyzed (Participants) | 93 | 103 | 196
    Open-label | 65.66 (20.867) | 68.01 (17.237) | 66.89 (19.033)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Test (6MWT)
Description: Change From Baseline in Distance Walked (meters) on the Six-Minute Walk Test by Visit
Time Frame: Baseline to 24 weeks
Population: All participants for whom 6MWT was measured
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Elamipretide: Double-blind Period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system
- Placebo: Double-Blind Period: Placebo comparator: 40 mg of placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
meters
  Week 4: number analyzed (Participants) | 108 | 105
  Week 4 | 16.243 (42.0071) | 7.811 (39.5737)
  Week 12: number analyzed (Participants) | 106 | 102
  Week 12 | 18.286 (47.7766) | 8.801 (52.1093)
  Week 24: number analyzed (Participants) | 100 | 102
  Week 24 | 15.330 (61.4860) | 17.386 (51.6956)

2. Primary Outcome: Total Fatigue Score on the on the Primary Mitochondrial Myopathy Symptom Assessment (PMMSA)
Description: Change from Baseline in Total fatigue score on the on the Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) by visit. Each individual item score ranges from 1 (none) to 4 (severe). The total fatigue score ranges from 4-16. Lower values represent a better outcome. The total fatigue score is the sum of question 1 through question 4 on the Primary Mitochondrial Myopathy Symptom Assessment.
Time Frame: Baseline to 24 weeks
Population: All participants for whom Total Fatigue Score (Q1 to Q4) Based on PMMSA by Visit was measured
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
score on a scale
  Week 4: number analyzed (Participants) | 106 | 105
  Week 4 | -1.01 (1.714) | -1.08 (1.865)
  Week 12: number analyzed (Participants) | 103 | 103
  Week 12 | -1.08 (1.775) | -1.26 (2.259)
  Week 24: number analyzed (Participants) | 98 | 101
  Week 24 | -1.18 (2.132) | -1.09 (2.443)

3. Secondary Outcome: Fatigue During Activities Score on the Primary Mitochondrial Disease Symptom Assessment (PMMSA).
Description: Change from baseline in Fatigue During Activities. Fatigue During Activities is the sum of question 2 (tiredness during activities) and question 4 (muscle weakness during activities.) The four response options are: 1=Not at all, 2=Mild, 3=Moderate, and 4=Severe. Raw scores for each subject range from 2-8. A lower score means a better outcome, with less fatigue. A higher score means a worse outcome, with more fatigue.
Time Frame: Baseline to 24 weeks
Population: All participants for whom Fatigue During Activities was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
score on a scale
  Week 4: number analyzed (Participants) | 106 | 105
  Week 4 | -0.48 (0.890) | -0.60 (0.998)
  Week 12: number analyzed (Participants) | 103 | 103
  Week 12 | -0.57 (0.923) | -0.67 (1.199)
  Week 24: number analyzed (Participants) | 98 | 101
  Week 24 | -0.64 (1.151) | -0.59 (1.360)

4. Secondary Outcome: Neuro-QoL Fatigue Activities of Daily Living
Description: Change From Baseline in Neuro-QoL Fatigue Activities of Daily Living by Visit. Each individual item score ranges from 1-5. Total raw score for the entire item bank ranges from 19-95. Raw scores will be calibrated using Item Response Theory Model. Lower values represent a better outcome. Individual items will be summed to calculate total scores.
Time Frame: Baseline to 24 weeks
Population: All participants for whom Change From Baseline in Neuro-QoL Fatigue Activities of Daily Living by Visit was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
score on a scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | -2.5 (5.33) | -2.7 (5.31)
  Week 12: number analyzed (Participants) | 106 | 104
  Week 12 | -2.9 (6.00) | -2.9 (5.13)
  Week 24: number analyzed (Participants) | 101 | 103
  Week 24 | -2.7 (6.06) | -2.1 (5.39)

5. Secondary Outcome: Change From Baseline in the Most Bothersome Symptom Score on the Primary Mitochondrial Myopathy Symptoms Assessment
Description: The item score rangers from 1 (none) to 4 (severe). Lower values represent a better outcome. The most bothersome score is the average of the identified most bothersome symptom of the Primary Mitochondrial Myopathy Symptom Assessment by each subject.
Time Frame: Baseline to 24 weeks
Population: All participants for whom Most Bothersome Symptom Score (PMMSA) by Visit was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
score on a scale
  Week 4: number analyzed (Participants) | 106 | 105
  Week 4 | -0.21 (0.492) | -0.24 (0.535)
  Week 12: number analyzed (Participants) | 103 | 103
  Week 12 | -0.24 (0.535) | -0.34 (0.656)
  Week 24: number analyzed (Participants) | 98 | 101
  Week 24 | -0.25 (0.618) | -0.30 (0.713)

6. Secondary Outcome: Neuro-QoL Fatigue Short Form Score
Description: Change From Baseline in Neuro-QoL Fatigue - Short Form: Total T-Scores by Visit. The Neuro-QoL Fatigue Short Form is comprised of the sum of the first 8 questions of the Neuro-QoL Item Bank v1.0 - Fatigue. Each question is scored as following: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, and 5=Always. The questions include: I felt exhausted, I felt that I had no energy, I felt fatigued, I was too tired to do my household chores, I was too tired to leave the house, I was frustrated by being too tired to do the things I wanted to do, I felt tired, and I had to limit my social activity because I was tired. T-scores are calculated from the short form scoring table provided by the instrument authors (Neuro-QoL User Manual, 2015). T-score distributions rescale raw scores into standardized scores with a mean of 50 and a standard deviation (SD) of 10. Change from baseline: Negative numbers mean less fatigue, better outcome, positive score means more fatigue, worse outcome.
Time Frame: 24 Weeks
Population: All participants for whom Neuro-QoL Fatigue Short Form Score T-scores were measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 109 | 109
score on a scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | -3.37 (5.077) | -2.89 (5.915)
  Week 12: number analyzed (Participants) | 106 | 104
  Week 12 | -3.43 (5.681) | -3.60 (5.614)
  Week 24: number analyzed (Participants) | 101 | 103
  Week 24 | -2.68 (5.769) | -2.61 (5.773)

ADVERSE EVENTS:
Time Frame: Double-blind period: 24 weeks and continued with Open-label period: up to 144 weeks.
Groups:
- Double-Blind Elamipretide: Double-blind period: elamipretide: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system, then elamipretide open-label treatment: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
- Double-Blind Placebo: Placebo SC daily
  Double-blind period: placebo comparator: Placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system. Open-label period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system.
- Open-Label Elamipretide: Double blind period: elamipretide: 40mg (0.5mL) of elamipretide administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system, then elamipretide open-label treatment: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system
- Open-Label Placebo: Double-blind period: placebo comparator: Placebo administered as once daily 0.5 mL subcutaneous injections for 24 weeks using the elamipretide delivery system. Open-label period: 40 mg of elamipretide administered as once daily 0.5 mL subcutaneous injections for up to 144 weeks using the elamipretide delivery system.
Arm/Group | Double-Blind Elamipretide | Double-Blind Placebo | Open-Label Elamipretide | Open-Label Placebo
All-Cause Mortality (participants affected / at risk) | 0/109 | 0/109 | 0/93 | 0/103
Serious Adverse Events (participants affected / at risk) | 5/109 | 3/109 | 12/93 | 9/103
Other Adverse Events (participants affected / at risk) | 107/109 | 83/109 | 88/93 | 102/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Elamipretide (N=109) | Double-Blind Placebo (N=109) | Open-Label Elamipretide (N=93) | Open-Label Placebo (N=103)
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Viral sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Lactic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Psychogenic seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery dissection (Cardiac disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
MELAS syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Vaginal laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Labile blood pressure (Vascular disorders) | 0 | 0 | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double-Blind Elamipretide (N=109) | Double-Blind Placebo (N=109) | Open-Label Elamipretide (N=93) | Open-Label Placebo (N=103)
Injection site erythema (General disorders) | 94 | 31 | 66 | 87
Injection site pruritus (General disorders) | 82 | 10 | 57 | 81
Injection site pain (General disorders) | 43 | 20 | 32 | 37
Injection site swelling (General disorders) | 42 | 7 | 29 | 20
Injection site induration (General disorders) | 31 | 6 | 25 | 41
injection site bruising (General disorders) | 9 | 18 | 5 | 15
injection site haemorrhage (General disorders) | 7 | 10 | 2 | 8
injection site urticaria (General disorders) | 14 | 0 | 12 | 8
injection site nodule (General disorders) | 11 | 2 | 8 | 8
injection site mass (General disorders) | 9 | 2 | 4 | 4
Fatigue (General disorders) | 4 | 4 | 4 | 4
injection site haematoma (General disorders) | 0 | 7 | 0 | 0
Pyrexia (General disorders) | 2 | 3 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 3 | 2
Injection site injury (General disorders) | 0 | 0 | 1 | 4
Upper respiratory tract Infection (Infections and infestations) | 7 | 7 | 7 | 7
Nasopharyngitis (Infections and infestations) | 8 | 2 | 6 | 2
Sinusitis (Infections and infestations) | 2 | 3 | 2 | 4
Headache (Nervous system disorders) | 8 | 4 | 5 | 6
Dizziness (Nervous system disorders) | 6 | 3 | 1 | 3
Nausea (Gastrointestinal disorders) | 5 | 8 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 9 | 3 | 6
Eosinophil count increased (Investigations) | 7 | 0 | 7 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 5
Fall (Injury, poisoning and procedural complications) | 6 | 3 | 8 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3 | 3
Influenza (Infections and infestations) | 0 | 0 | 2 | 2
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 4 | 1
Weight Decreased (Investigations) | 0 | 0 | 2 | 3
Blood glucose increased (Investigations) | 0 | 0 | 2 | 2
Blood lactic acid increased (Investigations) | 0 | 0 | 2 | 2
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 3
Migraine (Nervous system disorders) | 0 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 3 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 9
Hypertension (Vascular disorders) | 0 | 0 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/49/NCT03323749/Prot_001.pdf
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT03323749/SAP_002.pdf